CLINICAL TRIAL: NCT06014229
Title: Thermal Ablation of Benign Thyroid Nodules with Cryoablation
Brief Title: Cryoablation of Benign Thyroid Nodules: a Pilot Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5.712.194
Record Dates: First submitted 2023-08-22; First posted 2023-08-28 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-10

CONDITIONS: Benign Thyroid Nodule
MeSH Terms: interventions — Cryosurgery

STUDY DESIGN:
Intervention Model Description: pilot study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Cryoablation (Experimental): Device: Cryoablation Single session with an argon-based device; a V-probe 17-G applicator will be used for the treatments; gas release 100%; local anesthesia or moderate sedation or general anesthesia at discretion of the anesthesiology / interventional radiology team; benign thyroid nodules (two benign cytological examinations) measuring between 5 and 65 mL of volume and less than 40% of cystic component;
  Interventions: Device: cryoablation

INTERVENTIONS:
Device: cryoablation — Single session with an argon-based cryoablation device; an specific applicator will be used for the treatments; gas release 100% for cryoablation; local anesthesia or moderate sedation or general anesthesia at discretion of the anesthesiology / interventional radiology team; benign thyroid nodules (two benign cytological examinations) measuring between 5 and 65 mL of volume and less than 40% of cystic component;

SUMMARY:
This study will evaluate the clinical response and safety of ultrasound guided percutaneous cryoablation in the treatment of benign thyroid nodules as an alternative to the surgery. Ablation of functioning or non-functioning benign thyroid nodules with cryoablation will be directed to patients with symptomatic benign thyroid lesions (two benign cytological examinations) measuring between 5 and 65 mL of volume and less than 40% of cystic component; patients must present with serum free thyroxine (T4) and thyroid stimulating hormone (TSH) between the normal range values, with no signs of thyroiditis by serum antibodies over 100% of the standard values; calcitonin levels in the normal range values. Cryoablation will be directed to patients in a non-randomized fashion. Clinical, laboratorial and imaging monitoring will be performed in 12 months, including contrast-enhanced ultrasound when indicated, by 1, 3, 6 and 12 months.

DETAILED DESCRIPTION:
Palpable nodular thyroid disease is common in up to 6.4% of the population, and it becomes more common when the thyroid is examined by ultrasound. The vast majority of nodules are benign and, over time, do not change considerably in size. The main treatment indications for a euthyroid patient with a benign thyroid nodule that is not hyperfunctioning are compression of the trachea or esophagus, growth of the nodule, and recurrence of a cystic nodule after aspiration. Other indications for treatment are neck discomfort, cosmetic concern, and patient anxiety about the lump. The main therapeutic options are surgery (unilateral lobectomy) and treatment with thyroxine. Thermal ablative therapy has become a treatment option for solid thyroid lesions, with extensive reports in the medical literature on safety and efficacy with laser and radiofrequency devices, including long-term follow-up studies (10 years). There is no record in the medical literature of the use of cryoablation devices for the ablation of benign thyroid nodules, although they are used for the treatment of tumor lesions in different sites (hepatic, renal, pulmonary, bone and cervical lymph nodes).The objective of this research is to evaluate, in a pilot study, the safety and efficacy of cryoablation in the treatment of benign thyroid nodules.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Patients with solitary or dominant functioning or non-functioning thyroid nodules with two consecutive fine needle aspiration biopsy (FNAb)-proven benign in the last 12 months
* Thyroid nodules should be solid or almost solid (less than 40% of liquid component) with volume between 5 and 65 cc;
* Patients considered high surgical risk candidates or patients are eligible to surgery who are informed about the ablation therapy and prefers it instead surgery;
* Calcitonin, thyroglobulin or TSH serum levels in the normal range values

Exclusion Criteria:

* Age under 18 years
* Extensive goiter
* Predominantly cystic nodule with small solid remnant (less than 10%)
* Nodule volume > 65 cc
* TSH levels above the normal range
* Uncorrectable coagulopathy / impossibility to interrupt anticoagulants;
* Malignant or suspected malignant cytologic specimens;
* Pregnancy or breast-feeding;
* Anaplastic or poor-differentiated thyroid carcinoma;
* Partial thyroidectomy
* Asymptomatic patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-08-24 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
evaluation of technical feasibility | immediately after ablation
  Defined as the ability to puncture the nodule and perform the ablation as preoperatively planned.
2) Incidence of adverse events secondary to the treatment (safety and tolerability) of thermal ablation of benign thyroid nodules | up to 4 weeks after ablation
  Evaluation of minor and major complication rates, immediately after and 1 month after ablation [designed as a safety measure: yes]. The safety endpoint for this study is to evaluate the incidence and severity of the procedure or device-related adverse events, as reported by the CTCAE V5.2017.

SECONDARY OUTCOMES:
Evaluation of technical success | ultrasound examinations 1, 3, 6 and 12 months after ablation
  Technical success is defined as to achieve a nodular volume ablation of 50% at 12-month follow up compared to baseline. Nodule volume measurement is performed with the ellipsoid formula: length x width x depth x 0.524.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Freitas, MD, PhD, Principal Investigator — Instituto de Radiologia - Hospital das Clínicas da Universidade de São Paulo
Locations (1):
- University of Sao Paulo General Hospital, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No